CLINICAL TRIAL: NCT03633916
Title: Effects of a Classroom-based Sensitization Intervention on Demand for Mental Health Care Among School-going Adolescents in New Delhi, India: Study Protocol for a Stepped-wedge Cluster Randomized Controlled Trial
Brief Title: Impact of a Classroom-based Sensitization Intervention on Demand for Mental Health Care Among Adolescents in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sangath (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SANPRIDE_003
Record Dates: First submitted 2018-08-10; First posted 2018-08-16 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Help-Seeking Behavior
Keywords: adolescents; urban; school; demand for mental health care
MeSH Terms: conditions — Help-Seeking Behavior

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Classroom sensitization session (plus school-level sensitization activities)
  Interventions: Behavioral: Classroom sensitization session; Behavioral: School-level sensitization activities
- Control (Active Comparator): School-level sensitization activities only
  Interventions: Behavioral: School-level sensitization activities

INTERVENTIONS:
Behavioral: Classroom sensitization session — A one-off classroom information and engagement session will be delivered in addition to school-level sensitization activities. Individual classroom sessions will be conducted by a 'lay' counsellor with support from a researcher.
  The classroom session will start with a short animated video which provides age-appropriate information about types, causes, impacts and ways of coping with common mental health problems. The video will be followed by a guided group discussion, structured around a standardized script that builds on the topics covered in the video. In case of technical difficulties that may prevent the video from being shown, a flipchart based on still illustrations from the video will be used.
  At the end of the session, students will be handed a self-referral form which includes normalizing information and question-based prompts to assist with self-identification of mental health problems.
  Arms: Intervention
Behavioral: School-level sensitization activities — The control condition intervention will comprise sensitization activities conducted at the whole school level. These activities will include:
  1. Posters containing information about the school counselling program and referral pathways will be displayed in prominent locations at each school.
  2. A drop-box for student self-referral slips will be set up in a prominent location at each school.
  3. Information meetings with teachers and the principal will be conducted at each school from the beginning of the trial.

SUMMARY:
The primary objective of this embedded stepped-wedge, cluster randomized controlled trial is to evaluate the impact of a classroom sensitization (intervention condition), over and above the school-level sensitization activities (control condition), on referrals to a host trial (examining the effectiveness of a problem-solving intervention delivered by lay counsellors). The primary hypothesis is that the classroom-level sensitization intervention will be associated with a higher overall referral rate into the host trial (i.e. the proportion of adolescents referred as a function of the total sampling frame in each condition). The secondary hypotheses are that, compared with the control condition, the intervention condition will be associated with a greater proportion of referred students who meet eligibility criteria for inclusion in the host trial and a greater proportion of students who self-refer. We will also explore whether there are any differences between conditions in terms of the severity of total symptoms and symptom subtypes presented by referred adolescents.

DETAILED DESCRIPTION:
Background and rationale:

Schools are recommended as strategically important platform for improving young people's access to mental health care, including in low and middle- income countries (Patton et al., 2016). Along with a limited supply of effective treatments, low awareness about mental health problems and their treatment often act as barriers to help seeking in schools. Interventions to increase mental health literacy have been shown to increase the demand for mental health care among young people in a number of studies conducted worldwide, including in low-resource settings. However, the evidence is not conclusive as many of the existing studies are associated with a high risk of bias (Wei et al., 2013; Wei et al., 2015; Kutcher et al., 2016).

Formative research in Government-run secondary schools in New Delhi, India indicated that mental health services were non-existent and adolescents had limited knowledge about mental health care. The investigators have therefore developed sensitization activities to promote referral to, and uptake of, a newly developed school counselling service. These sensitization activities have been designed for implementation at both whole school and classroom-levels, and are intended to be delivered by non-specialist counsellors. The additional resource investment in classroom-level sensitization activities may be justified if this component leads to significantly greater levels of demand. This trial therefore seeks to evaluate the additional impact of the classroom sensitization session on demand for school counselling in New Delhi.

This study is part of a larger research program called PRIDE (PRemIum for aDolEscents). The overall goal is to develop and evaluate a trans-diagnostic, stepped-care intervention targeting common mental disorders in school-going adolescents in India. The PRIDE intervention architecture involves two sequential psychological treatments of incremental intensity. The first step is a brief problem-solving intervention delivered by lay counsellors. Adolescents with enduring mental health problems are referred to a higher intensity trans-diagnostic treatment delivered by psychologists.

The trial described here is embedded within a host trial that is testing the effectiveness of the low-intensity problem-solving intervention. The embedded trial will evaluate the impact of the classroom sensitization activities over and above the school-level activities on referral rates generated for the host trial.

Study design and setting:

An embedded recruitment trial will apply a stepped-wedge, cluster (class)-randomized controlled design in 70 classes across six Government-run secondary schools in New Delhi.

Eligibility criteria: Please see section on eligibility.

Interventions: Please see section on Intervention arms.

Outcomes: Please see section on outcome measures.

Trial scheme:

The trial will be conducted over 12 weeks and recruit 70 classes. The referral outcomes for the students will be reported every four weeks across these classes. As each class has an average enrollment of 50, the study will follow around 3400 students for the entire trial duration of 12 weeks.

Each class will switch over from the control condition to the intervention condition at 4-week intervals (excluding holidays and exam breaks), over 2 steps. During the first 4-week period, only school-level sensitization activities will be implemented. In the next 4-week period (first step), 35 randomly selected classes (sequence 1) will receive the classroom sensitization intervention. In the final 4-week period (second step), the remaining 35 classes (sequence 2) will receive the classroom sensitization intervention. Schedules for sensitization in the allocated classes will be shared with the schools in advance to ensure access.

Power calculation:

We based our power calculation on a within-period comparison for a stepped wedge design (Thompson et al., 2018) using Stata package "clustersampsi". Based on pilot data, we anticipated referral rates of 5% and 15% on the control and intervention conditions respectively, with an intra-cluster correlation coefficient (ICC) of 0.124. Using these parameters, a sample size of 70 classes (average class size of 50 students) will have 92% power to detect a difference of 10 percentage points (treating the outcome as a binomial variable), at a significance level of 0.05.

Data collection:

The primary outcome (referral rate) will be collated from referral logs maintained by researchers in each school. Referral data will be aggregated over each 4-week period. Secondary outcomes pertaining to the eligibility and clinical characteristics of students referred to the host trial will be derived from the Strengths and Difficulties Questionnaire (SDQ; Goodman et al., 2000).

Statistical analysis:

The baseline characteristics of the participating 70 classes, including class size and gender composition, will be described and assessed for any systematic differences across the two sequences. The primary outcome will be analyzed using generalized estimating equations (GEE) with robust standard errors. GEE is a recommended method for analysis of stepped-wedge cluster randomized controlled trials, providing population-averaged effects of exposure across trial conditions (Barker et al., 2016). GEE allows for longitudinal data analysis without resorting to fully specified random effect models and can be applied to both continuous and categorical outcomes (Liang and Zeger, 1986). It provides both parameter estimates and standard errors that are corrected for clustering of data and are consistent despite misspecifications in the correlation structure. For this trial, the clustering of data will be specified at the class level. Analysis of the secondary and exploratory outcomes will also be undertaken using the GEE method. Sensitivity analysis will be conducted using a 'within-period comparison' of data from the second period only (Thompson et al., 2018). No interim analysis will be undertaken.

Process evaluation:

We will undertake descriptive analysis of quantitative process data in order to explore potential sources of variation in the implementation of intervention procedures.

ELIGIBILITY:
CLASSROOM CLUSTERS

Inclusion criteria:

* Classes from grades 9-12 in the six collaborating schools.

Exclusion criteria:

* Classes that have received classroom sensitization sessions during earlier pilot work.

ADOLESCENT PARTICIPANTS

Inclusion criteria:

* Enrolled as a student in grades 9-12 (aged 13-20 years) at one of the collaborating schools
* Adolescent willing and able to consent for participation in the research

Exclusion criteria:

* Adolescent not proficient in written and spoken Hindi, as needed to participate fully in study procedures
* Adolescent needing urgent medical or mental health care

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 835 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Referral rate into the host trial | 4 weeks
  The referral rate will be calculated as the number of referred students from a given condition divided by the total number of students in corresponding classes. This will be calculated from researchers' referral logs. Referrals will be recorded continuously and reported for each 4 weeks' time period, for the total study duration of 12 weeks.

SECONDARY OUTCOMES:
Eligibility rate | 4 weeks
  Eligibility rate is defined as the proportion of referred participants meeting eligibility criteria for the host trial, as a function of the number of referred adolescents in a given condition. Host trial eligibility criteria are as follows: (i) Total Difficulties score on the adolescent-reported Strengths and Difficulties Questionnaire (SDQ; Goodman et al, 2000) >/= 19 for boys & >/= 20 for girls; (ii) SDQ Impact Supplement score of >/=2; and (iii) chronicity of mental health problems for >/= 1 month. Referred students will complete the SDQ as part of the host trial's screening assessment, within 7 working days of the referral date. Eligibility rate will be calculated for each of the 4-week time periods and reported for the entire study duration of 12 weeks.
Self-referral rate | 4 weeks
  Self-referral rate is defined as the proportion of referrals which are self-initiated as a function of the number of referred adolescents in a given condition. Self-referral rate will be calculated for each of the 4-week time periods and reported for the entire study duration of 12 weeks, based on data from researchers' referral logs

OTHER OUTCOMES:
Severity of mental health symptoms | 4 weeks
  Severity of mental health symptoms will be assessed as an exploratory outcome for students referred across the control and intervention conditions. The SDQ total difficulties score will be used to assess the severity of mental health symptoms. It is calculated by adding the scores of all the SDQ sub-scales except the pro-social scale.
Severity of symptom subtypes | 4 weeks
  Internalizing and externalizing symptom subtypes will be assessed as an exploratory outcome for the students referred across the control and intervention conditions. The externalising symptoms score is calculated as the sum of the conduct and hyperactivity sub-scales. The internalising symptoms score is calculated as the sum of the emotional and peer relationship problem sub-scales.

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Patel, MRCPsych PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Sangath, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data along with data dictionaries will be shared with other researchers after 12 months of completion of the trial. Data pertaining to the interventions received and outcomes will be shared upon reasonable requests made to the PI and in accordance with the guidelines of the sponsor, collaborating institutions and funder of the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after completion of trial.
Access Criteria: Access to data will be granted to researchers after review of requests by PI and in accordance with the guidelines of the sponsor, collaborating institutions and funder of the study.
URL: http://datacompass.lshtm.ac.uk/

REFERENCES:
- [Background] Patton GC, Sawyer SM, Santelli JS, Ross DA, Afifi R, Allen NB, Arora M, Azzopardi P, Baldwin W, Bonell C, Kakuma R, Kennedy E, Mahon J, McGovern T, Mokdad AH, Patel V, Petroni S, Reavley N, Taiwo K, Waldfogel J, Wickremarathne D, Barroso C, Bhutta Z, Fatusi AO, Mattoo A, Diers J, Fang J, Ferguson J, Ssewamala F, Viner RM. Our future: a Lancet commission on adolescent health and wellbeing. Lancet. 2016 Jun 11;387(10036):2423-78. doi: 10.1016/S0140-6736(16)00579-1. Epub 2016 May 9. No abstract available. PMID 27174304
- [Background] Wei Y, McGrath PJ, Hayden J, Kutcher S. Mental health literacy measures evaluating knowledge, attitudes and help-seeking: a scoping review. BMC Psychiatry. 2015 Nov 17;15:291. doi: 10.1186/s12888-015-0681-9. PMID 26576680
- [Background] Kutcher S, Wei Y, Costa S, Gusmao R, Skokauskas N, Sourander A. Enhancing mental health literacy in young people. Eur Child Adolesc Psychiatry. 2016 Jun;25(6):567-9. doi: 10.1007/s00787-016-0867-9. No abstract available. PMID 27236662
- [Background] Wei Y, Hayden JA, Kutcher S, Zygmunt A, McGrath P. The effectiveness of school mental health literacy programs to address knowledge, attitudes and help seeking among youth. Early Interv Psychiatry. 2013 May;7(2):109-21. doi: 10.1111/eip.12010. Epub 2013 Jan 24. PMID 23343220
- [Background] Goodman R, Ford T, Simmons H, Gatward R, Meltzer H. Using the Strengths and Difficulties Questionnaire (SDQ) to screen for child psychiatric disorders in a community sample. Br J Psychiatry. 2000 Dec;177:534-9. doi: 10.1192/bjp.177.6.534. PMID 11102329
- [Background] Thompson JA, Davey C, Fielding K, Hargreaves JR, Hayes RJ. Robust analysis of stepped wedge trials using cluster-level summaries within periods. Stat Med. 2018 Jul 20;37(16):2487-2500. doi: 10.1002/sim.7668. Epub 2018 Apr 10. PMID 29635789
- [Background] Barker D, McElduff P, D'Este C, Campbell MJ. Stepped wedge cluster randomised trials: a review of the statistical methodology used and available. BMC Med Res Methodol. 2016 Jun 6;16:69. doi: 10.1186/s12874-016-0176-5. PMID 27267471
- [Background] Liang K-Y, Zeger SL. Longitudinal data analysis using generalized linear models. Biometrika. 1986;73(1):13-22.
- [Derived] Parikh R, Hoogendoorn A, Michelson D, Ruwaard J, Sharma R, Bhat B, Malik K, Sahu R, Cuijpers P, Patel V. Increasing demand for school counselling through a lay counsellor-delivered classroom sensitisation intervention: a stepped-wedge cluster randomised controlled trial in New Delhi, India. BMJ Glob Health. 2021 Jun;6(6):e003902. doi: 10.1136/bmjgh-2020-003902. PMID 34172486
- [Derived] Parikh R, Michelson D, Malik K, Shinde S, Weiss HA, Hoogendoorn A, Ruwaard J, Krishna M, Sharma R, Bhat B, Sahu R, Mathur S, Sudhir P, King M, Cuijpers P, Chorpita BF, Fairburn CG, Patel V. The effectiveness of a low-intensity problem-solving intervention for common adolescent mental health problems in New Delhi, India: protocol for a school-based, individually randomized controlled trial with an embedded stepped-wedge, cluster randomized controlled recruitment trial. Trials. 2019 Sep 18;20(1):568. doi: 10.1186/s13063-019-3573-3. PMID 31533783

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT03633916/SAP_000.pdf